CLINICAL TRIAL: NCT07295054
Title: A Double-blind Placebo-controlled Randomized Controlled Trial (RCT) of 3 mL Inhaled Methoxyflurane for Intrauterine Device (IUD) Insertion
Brief Title: 3 mL Inhaled Methoxyflurane for Intrauterine Device (IUD) Insertion
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-0056-B
Record Dates: First submitted 2025-11-27; First posted 2025-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: IUD
Keywords: Methoxyflurane; Penthrox
MeSH Terms: interventions — Methoxyflurane; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study is designed as a double-blind, placebo-controlled randomized controlled trial (RCT) conducted at The Bay Centre for Birth Control Clinic at Women's College Hospital (WCH). The intervention will occur over a single study visit, with data collected at baseline, immediately prior to the procedure, and following the procedure using quantitative survey instruments. Participant recruitment is planned over an 18-month period.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: As noted above, only the individual preparing the intervention will be aware of allocation assignment. The participant, IUD provider, anesthesia provider and outcomes assessors will be blinded to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will receive a Penthrox inhaler containing 3 mL of methoxyflurane. Before speculum insertion, they will take intermittent inhalations every 30-60 seconds (6-10 breaths), following monograph instructions. They may continue self-administering the inhaler as needed during the procedure.
  Interventions: Drug: Penthrox
- Placebo Group (Placebo Comparator): Participants will receive an identical-looking inhaler containing 3 mL of normal saline. To maintain blinding, a drop of methoxyflurane will be placed on the outside of the device, which has no analgesic effect. Before speculum insertion, participants will take intermittent inhalations every 30-60 seconds (6-10 breaths), following monograph-style instructions, and may continue self-administering as needed during the procedure.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Penthrox — 3 mL of Methoxyflurane via a handheld inhaler
  Other Names: methoxyflurane
  Arms: Intervention Group
Drug: Saline — 3 mL of Normal Saline via an identical placebo handheld inhaler
  Arms: Placebo Group

SUMMARY:
Intrauterine device (IUD) insertion is a common contraceptive procedure often associated with moderate to severe pain, particularly among nulliparous individuals. Current pain management strategies, such as over-the-counter analgesics, are frequently inadequate. Methoxyflurane, a short-acting, self-administered inhaled analgesic, has been shown to provide rapid and effective pain relief in acute and procedural settings. This study aims to evaluate whether 3 mL of inhaled Methoxyflurane (via Penthrox inhaler) improves patient satisfaction by reducing pain and anxiety during IUD insertion.

DETAILED DESCRIPTION:
Methoxyflurane is a short-acting, self-administered inhaled analgesic that has demonstrated rapid and effective pain relief in acute trauma, emergency, and procedural settings. It is non-narcotic, allows patients to control dosing, and does not require intravenous access or prolonged recovery, making it suitable for short outpatient procedures. Existing studies indicate that Methoxyflurane provides faster onset of pain relief compared to standard analgesics, is generally well-tolerated, and has only transient, non-serious adverse effects such as dizziness or headache.

This study aims to evaluate the efficacy of 3 mL of inhaled Methoxyflurane, delivered via Penthrox inhaler, in reducing pain and anxiety during IUD insertion. The primary objective is to assess patient satisfaction with pain management. Secondary outcomes include procedural pain scores, anxiety levels, and the incidence of adverse events. This trial seeks to provide evidence for an effective, safe, and patient-centered approach to pain management during IUD insertion, potentially improving patient experience and access to long-acting contraceptive options.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a uterus.
2. Ages 18 to 55 years.
3. Undergoing any intrauterine device (IUD) insertion.
4. English-speaking participants.
5. Ability to use an inhaler device.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Confirmed pregnancy.
3. Use of pain medication other than NSAIDs or acetaminophen (e.g., opioids, benzodiazepines, muscle relaxants) within 24 hours prior to the intervention.
4. Use of cannabis within 24 hours prior to the intervention.
5. Administration of misoprostol within 24 hours prior to the intervention.
6. Altered level of consciousness due to any cause, including head injury, drugs, or alcohol.
7. History of severe adverse reactions to Penthrox (methoxyflurane) or other halogenated anesthetic agents, or to any ingredient in the formulation (including non-medicinal ingredients or container components).
8. Anatomical variance, such as distorted uterine cavity, bicornuate uterus, uterus didelphys, or cervical stenosis.
9. Clinically significant renal and/or liver impairment.
10. Known or genetic susceptibility to malignant hyperthermia.
11. Clinically evident hemodynamic or cardiovascular instability, or respiratory depression.
12. Not NPO according to hospital guidelines.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Procedural pain intensity | 20 minutes after post-procedure
  Patient-reported pain will be measured using the Numeric Rating Scale (NRS), a validated tool in which participants rate their pain intensity on a scale from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Patient-centered measure of satisfaction with procedural sedation | 20 minutes after post procedure
  PROcedural Sedation Assessment Survey (PROSAS)
Patient satisfaction with pain management | Baseline before procedure
  Pain Catastrophizing Scale (PCS) Purpose: To measure the extent to which individuals magnify, ruminate about, or feel helpless in response to pain.
  Structure:
  13 items rated on a 5-point Likert scale (0 = "not at all" to 4 = "all the time").
  Items are grouped into three subscales:
  Rumination - Focused on the inability to stop thinking about pain. Magnification - Exaggeration of the threat value of pain. Helplessness - Perceived inability to manage pain.
  Scoring:
  Total PCS score ranges from 0 to 52. Higher scores indicate greater pain catastrophizing. Subscale scores can also be calculated for more nuanced insights.
Patient distress | Pre-procedure and post procedure 0,20 minutes and 24 hours.
  Faces Anxiety Scale Faces are assigned numerical values (e.g., 0-5 or 0-10). Higher scores indicate greater anxiety.
Patient Anxiety | Pre-procedure and post procedure 0,20 minutes and 24 hours.
  State-Trait Anxiety Inventory (STAI)
  Structure:
  40 items in total:
  20 items for State Anxiety (S-Anxiety) 20 items for Trait Anxiety (T-Anxiety)
  Respondents rate items on a 4-point Likert scale:
  For State Anxiety: 1 = "Not at all" to 4 = "Very much so" For Trait Anxiety: 1 = "Almost never" to 4 = "Almost always"
  Scoring:
  Each subscale (State and Trait) is scored separately. Higher scores indicate higher levels of anxiety. Scores can be used to track changes over time or to compare anxiety levels across groups.
Recall peak pain during procedure | 0 minutes after post procedure
  Patient-reported pain will be measured using the Numeric Rating Scale (NRS), a validated tool in which participants rate their pain intensity on a scale from 0 (no pain) to 10 (worst imaginable pain).
Provider-centered measure of satisfaction with procedural sedation | 20 minutes after post procedure
  PROcedural Sedation Assessment Survey (PROSAS)
Assess the effectiveness of blinding | 20 minutes after post procedure
  Bang Blinding Index (BBI)- Patient, Assessor and Anesthesia provider
Symptom Reporting / Emergency Visits | 24 hours after post procedure
  Adverse Events recording
Patient Satisfaction with Pain Management | 20 minutes after post procedure
  Patient-reported satisfaction will be measured on a 5-point scale ranging from 0 (not satisfied) to 10 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Scott, NP, Principal Investigator — Women's College Hospital